CLINICAL TRIAL: NCT03240341
Title: Influence of PARAmedical Interventions on Patient ACTivation in the Cancer Care Pathway
Acronym: PARACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Hôpital Privé de la Loire (Unknown); Centre Hospitalier Emile Roux (Other); Clinique de l'infirmerie protestante de Lyon (Ambiguous); Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-01; 2017-A00235-48 (Other: ANSM)
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Activation Measure (PAM) (Experimental): completion of the PAM questionnaire
  Interventions: Behavioral: Patient Activation Measure Questionnaire

INTERVENTIONS:
Behavioral: Patient Activation Measure Questionnaire — Measure the level of patient engagement in cancer care pathway

SUMMARY:
The aim is to implement the Patient Activation Measure in paramedical practices as a tool to measure activation of patients in cancer care

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Cancer patient with an estimated life expectancy of at least one year
* Patient requiring immunotherapy or intravenous chemotherapy for any cancer according to the decision of the Multidisciplinary Consultation Meeting
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Refusal to participate, protected adult patient under guardianship.
* Patient disability to understand the course of the study
* Patient with documented history of cognitive or psychiatric disorders.
* Patient not understanding French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure Questionnaire | 12 month

SECONDARY OUTCOMES:
Patient Activation Measure Questionnaire | 6 and 12 months
Visual Analog Scale for confidence level measurement about treatment | 6 and 12 months
Anxiety and Depression HAD Questionnaire | 6 and 12 months
REALM Health Literacy Test | 6 and 12 months
Quality of Life Questionnaire EQ-5D | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fournel, MD, Principal Investigator — CHU de Saint-Etienne
Locations (6):
- France (6):
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Clinique de l'infirmerie protestante de Lyon, Lyon
  - Centre Hospitalier de Roanne, Roanne
  - CHU de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verot E, Bouleftour W, Macron C, Rivoirard R, Chauvin F. Effect of PARACT (PARAmedical Interventions on Patient ACTivation) on the Cancer Care Pathway: Protocol for Implementation of the Patient Activation Measure-13 Item (PAM-13) Version. JMIR Res Protoc. 2020 Dec 8;9(12):e17485. doi: 10.2196/17485. PMID 33289495